CLINICAL TRIAL: NCT04575675
Title: Effects of Dapagliflozin on Hypotensive Patients With Depressed Left Ventricular Ejection Fraction After Sacubitril/Valsartan Therapy
Brief Title: Dapagliflozin on Hypotensive Heart Failure Patients After Sacubitril/Valsartan Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Hung-Yu Chang, Attending Physician, Cheng-Hsin General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChenghsinGH
Record Dates: First submitted 2020-08-26; First posted 2020-10-05 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Hypotension; Heart Failure
Keywords: Heart failure; Dapagliflozin; Sacubitril/valsartan
MeSH Terms: conditions — Hypotension; Heart Failure | interventions — dapagliflozin; sacubitril and valsartan sodium hydrate drug combination; Adrenergic beta-Antagonists; Bisoprolol; Nebivolol; Carvedilol; Mineralocorticoid Receptor Antagonists; Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin with standard-of-care therapies for heart failure, including sacubitril/valsartan, beta-blocker, MRA, ICD and CRT
  Interventions: Drug: Dapagliflozin; Drug: Sacubitril-Valsartan; Drug: Beta blocker; Drug: Mineralocorticoid Receptor Antagonist; Device: Cardiac resynchronization therapy and/or implantable cardioverter defibrillator
- Standard of care (Placebo Comparator): Standard-of-care therapies for heart failure, including sacubitril/valsartan, beta-blocker, MRA, ICD and CRT
  Interventions: Drug: Sacubitril-Valsartan; Drug: Beta blocker; Drug: Mineralocorticoid Receptor Antagonist; Device: Cardiac resynchronization therapy and/or implantable cardioverter defibrillator

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10mg once daily
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Sacubitril-Valsartan — Sacubitril-Valsartan, maximal tolerated dosage
  Other Names: Entresto
Drug: Beta blocker — Cardio-selective beta-blocker, including carvedilol, bisoprolol, metoprolol or nebivolol
  Other Names: Concor, Betaloc zok, Nebilet, Carvedilol
Drug: Mineralocorticoid Receptor Antagonist — Mineralocorticoid receptor antagonist, including spironolactone or eplerenone
  Other Names: Aldactin, Inspra
Device: Cardiac resynchronization therapy and/or implantable cardioverter defibrillator — CRT-P, CRT-D or ICD if clinically indicated

SUMMARY:
The DAPA-HF trial demonstrated that dapagliflozin was able to reduce the risk of worsening heart failure events and cardiovascular death comparing to placebo in patients with reduced ejection fraction further to standard of care. However, hypotensive patients who generally have higher risks comparing to normotensive patients, were under represented in the DAPA-HF. The investigators aimed to evaluate clinical effects of dapagliflozin on hypotensive heart failure patients receiving chronic sacubitril/valsartan treatment.

DETAILED DESCRIPTION:
The DAPA-HF trial demonstrated that dapagliflozin was able to reduce the risk of worsening heart failure (HF) events and cardiovascular death comparing to placebo in patients with reduced ejection fraction further to standard of care. However, hypotensive patients who generally have higher risks comparing to normotensive patients, were under represented in the DAPA-HF. The investigators aimed to evaluate clinical effects of dapagliflozin on hypotensive HFrEF patients receiving chronic sacubitril/valsartan (Sal/Val) treatment.

This is an investigator-initiated, interventional, prospective. open-label study. The inclusion criteria were (1) chronic symptomatic HF with New York Heart Association (NYHA) class II-IV and LVEF less than 40%, (2) treatment with stable and maximal tolerable dose of Sac/Val, beta-blocker with or without mineralocorticoid receptor antagonist (MRA), (3) 6-minute walking-distance (6MWD)≥ 100meters and ≤425 meters at enrollment, (4) systolic blood pressure ≤100 mmHg at enrollment. The exclusion criteria were (1) type 1 diabetes mellitus, (2) patients previously treated with any sodium glucose co-transporter 2 inhibitor (SGLT2i).

After applying the inclusion and exclusion criteria, if the participants had type 2 diabetes mellitus, the participants will receive dapagliflozin 10mg daily directly. If the participants did not have history of diabetes mellitus, the participants will be allocated to either receiving dapagliflozin 10mg daily or receiving standard heart failure treatment without dapagliflozin.

Vital signs and laboratory tests were examined at baseline, 2-week, 4-week and 12-week. Six-minute-walking-test, five-level EuroQol five dimensions (EQ-5D-5L) questionnaire and visual analogue scale (VAS) were collected at baseline and at 12-week.

ELIGIBILITY:
Inclusion Criteria:

* chronic symptomatic HF with New York Heart Association (NYHA) class II-IV and left ventricular ejection fraction (LVEF) less than 40%
* treatment with stable and maximal tolerable dose of Sac/Val, beta-blocker with or without mineralocorticoid receptor antagonist
* 6-minute walking-distance (6MWD)≥ 100meters and ≤425 meters at enrollment
* systolic blood pressure ≤100 mmHg at enrollment

Exclusion Criteria:

* hemodialysis
* severe co-morbidities with life expectancy less than 1 year
* type 1 diabetes mellitus
* ever treated with any type of sodium glucose cotransporter 2 inhibitor (SGLT2i)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
6-minute walking distance | 12 weeks
  Measuring walking distance within 6 minutes

SECONDARY OUTCOMES:
EQ-5D-5L | 12 weeks
  Measuring health status. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.This version of EQ-5D has five-level scale, The number of levels of severity was classified into: having no problems, having slight problems, having moderate problems, having severe problems and being unable to do/having extreme problems. This version can define 3,125 (5x5x5x5x5) different health states.
  Valuation of the EQ-5D-5L was then calcuated by the Taiwanese hybrid model, range from -1.0259 to 1. [PLoS One 13(12):e0209344]. Higher score indicates better health status.
EQ-Visual analogue scale (EQ-VAS) | 12 weeks
  Evaluating the participants' overall health status. The participant would be asked to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. There are notes at the both ends of the scale that the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yu Chang, MD, Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No